CLINICAL TRIAL: NCT04254354
Title: Masculinizing Testosterone Treatment and Effects on Preclinical Cardiovascular Disease, Muscle Strength and Power, Aggression, Physical Fitness and Respiratory Function in Transgender Men,Body Identity Clinic (BIC)
Brief Title: Transgender Men, Non-binary Persons and Testosterone Treatment BODY IDENTITY CLINIC
Status: Recruiting | Type: Observational
Sponsor: Marianne Andersen (Other)
Responsible Party: Sponsor-Investigator, Marianne Andersen, Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Other Study IDs: BICTX01
Record Dates: First submitted 2020-01-21; First posted 2020-02-05 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Transgenderism
MeSH Terms: conditions — Transsexualism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, hair
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- transgender men: no intervention

SUMMARY:
The aim of this study is to investigate transgender men and non-binary persons before and during testosterone treatment. The study will focus on:

* Cardiovascular status
* Muscle strenght and power
* Aggression and quality of life
* Cardiac and respiratory function

DETAILED DESCRIPTION:
Introduction: The number of individuals with gender dysphoria seeking gender-affirming treatment is increasing. The short- and long-term effects of masculinizing treatment with testosterone are debated as serum testosterone increase up to 20-fold compared to cisgender women. We hypothesize that, testosterone treatment is associated with non-calcified coronary plaque (NCP) development in transgender men.

Methods and analyses: Prospective, single-center, observational cohort study at the Body Identity Clinic (BIC), Odense University Hospital, Denmark, where all investigations are performed at inclusion and after 1, 3, 5 and 10 years of testosterone therapy.

Ethics and dissemination: The Regional Committees on Health Research Ethics for Southern Denmark (S-20190108) and the Danish Data Protection Agency approved the study (19/27572). Signed informed consent will be obtained from all participants. All findings will be published in peer-reviewed journals or at scientific conferences.

ELIGIBILITY:
Inclusion Criteria:

Transgender men

Exclusion Criteria:

none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Persons assigned female at birth (+18 years) that either use or want to use testosterone with the purpose of undergoing gender transformation. -
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-03-03 (Actual); Primary Completion 2044-01-01 (Estimated); Study Completion 2044-01-01 (Estimated)

PRIMARY OUTCOMES:
Effect of testosterone on devellopment of plaques in the heart | 10 years
  Estimated directly by CCTA, at start, (1 year for early included participants) 5 and 10 years

SECONDARY OUTCOMES:
Calcium score | 10 years
  CCTA
Change in muscle strength and power | 10 years
  Estimated by low row and accelometer at start, 1, 3, 5, 10 years
Effect of transgender treatment on quality of life | 10 years
  Estimated by quality of life questionnaire (SF36) at start, 1, 3, 5 and 10 years
Effect of transgender treatment on aggression | 10 years
  Estimated by aggression questionnaire at start, 1, 3, 5 and 10 years
Changes in maximal oxygen consumption during transgender treatment | 10 years
  Estimated by test og maximal oxygen consumption (vo2max) at start, 1, 3, 5 and 10 years
Heart function | 10 years
  Ejection fraction and left ventricular muscle mass are measured by echocardiography at start,(1 for early included participants) 5 and 10 years
Respiratory function | 10 years
  Forced Expiratory Volume in the first second and forced vital capacity estimated by spirometry at start, 1, 3, 5 and 10 years
Levels of testosterone, estradiol and cortisol | 10 years
  Measured in serum by LCMS/MS
circulating markers of inflammation | 10 years
  CRP in blood samples
circulating markers of cardiovascular risk | 10 years
  Lipids, SuPAR in blood samples
Assessment of cortisol/cortisone | 10 years
  measured in urine and hair samples by LCMS/MS
Change in lean body mass | 10 years
  Estimated by dual x-ray absorptiometry at start, 1, 3, 5 and 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Andersen, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lehmann Christensen L, Glintborg D, Taulbjerg Kristensen T, Diederichsen A, T'Sjoen G, Frystyk J, Skovsager Andersen M. Masculinising testosterone treatment and effects on preclinical cardiovascular disease, muscle strength and power, aggression, physical fitness and respiratory function in transgender men: protocol for a 10-year, prospective, observational cohort study in Denmark at the Body Identity Clinic (BIC). BMJ Open. 2020 Dec 29;10(12):e045714. doi: 10.1136/bmjopen-2020-045714. PMID 33376186